CLINICAL TRIAL: NCT04913831
Title: Effects of Cerebrolysin on Level of Consciousness and Brain Metabolism in Disorder of Consciousness After Stroke: Single Center Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2021-0085
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebrolysin (Experimental)
  Interventions: Drug: Cerebrolysin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin 20ml + physiological saline 80ml, 8-35 days, once/day, intravenous administration
  Arms: Cerebrolysin
Drug: Placebo — physiological saline 100ml, 8-35 days, once/day, intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the effect of stroke on post-stroke level of consciousness through a double-blind, placebo-controlled, randomized study design. And Brain 18F-FDG PET was used to reveal the mechanism of recovery after cerebrolysin administration.

Thirty patients with chronic stroke patients with minimal consciousness (MCS) or vegetative human (VS) level of consciousness disorder in the revised coma recovery scale were enrolled. Thirty patients were randomly divided into a Cerebrolysin group and a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke patients
* Stroke with CT or MRI diagnosis
* Chronic patients with more than 3 months of stroke onset
* Patients with vegetative status or minimal consciousness (Coma Recovery Scale -revised: CRS-R)
* Age: 19 to 90 years old
* A person who voluntarily consents to the clinical trial in writing by the principal or legal representative

Exclusion Criteria:

* In case of contraindications, including allergies to cerebrolysin
* Patients with contraindications to PET
* Progressive or unstable stroke
* In case of accompanying serious neurogenic disease
* Major depressive disorder, schizophrenia, bipolar disorder, dementia, and other serious psychiatric diseases.
* History of alcohol or other drug addiction within 3 years of onset
* In case of accompanying serious liver, kidney, heart, or respiratory disease
* If you have the following medical abnormalities (Total serum bilirubin> 4 mg/dL, alkaline phosphatase> 250 U/L, SGOT/AST> 150 U/L, SGPT/ALT> 150 U/L, or creatinine) > 3.5 mg/dL)
* In case of having a medical disease that is less than 1 year old
* During pregnancy or lactation
* Participating in other therapeutic research

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
CRS-R (JFK Coma recovery scale-revised) | up to 11 weeks
  It is a test that analyzes a total of six functions of hearing, vision, movement, speech, communication, and arousal by item to determine the improvement in the level of consciousness of patients with decreased consciousness. These items are scored to determine whether they are in a minimally conscious state (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No